CLINICAL TRIAL: NCT03558516
Title: The Effect of Magnesium Sulphate on Intraoperative Blood Loss in Meningioma Patient Undergoing Craniotomy With Tumor Removal
Brief Title: Magnesium and Intraoperative Blood Loss in Meningioma Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: SI 259/2018
Record Dates: First submitted 2018-05-16; First posted 2018-06-15 (Actual); Results first posted 2020-07-13 (Actual); Last update posted 2020-07-13 (Actual); Status verified 2020-06

CONDITIONS: Meningioma
Keywords: Meningioma; Magnesium; Montreal cognitive assessment; blood loss; controlled hypotension; blood transfusion; neuroprotective; anesthesia
MeSH Terms: conditions — Meningioma; Hemorrhage

STUDY DESIGN:
Intervention Model Description: We compare intraoperative blood loss in two group between the magnesium (study group) and 0.9% sodium chloride group (control group)
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: The study drug will prepared by the investigator in the same character and amount. So the patient and care provider will not know the study drug is magnesium or 0.9% sodium chloride.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Magnesium group (Experimental): The patient will receive magnesium sulfate injection 40 mg/kg infuse over 30 min started at skin incision and continuous drip 10 mg/kg/hr until the dura is closed
  Interventions: Drug: Magnesium group
- Normal saline group (Placebo Comparator): The patient will receive 0.9% sodium chloride the same amount of magnesium sulphate infuse over 30 min started at skin incision and continuous drip until the dura is closed
  Interventions: Drug: Normal saline group

INTERVENTIONS:
Drug: Magnesium group — We will dilute magnesium 6 gram with 0.9% sodium chloride to 30 ml. The patient will receive magnesium sulfate 40 mg/kg infuse over 30 min started at skin incision and continuous drip 10 mg/kg/hr until the dura is closed. Anesthesia is standardized with propofol, fentanyl, cisatracurium and sevoflurane. Vasopressor or antihypertensive drug are used to control hemodynamics.
  Other Names: Mg
  Arms: Magnesium group
Drug: Normal saline group — The patient will receive 0.9% sodium chloride the same amount of magnesium sulphate infuse over 30 min started at skin incision and continuous drip until the dura is closed. Anesthesia is standardized with propofol, fentanyl, cisatracurium and sevoflurane. Vasopressor or antihypertensive drug are used to control hemodynamics.
  Other Names: NSS
  Arms: Normal saline group

SUMMARY:
Meningioma is the most common central nervous system tumor and craniotomy with tumor removal was associated with moderate blood loss and blood transfusion. Magnesium has hypotensive effect and probably reduce intraoperative blood loss. Whether or not magnesium sulphate can reduce intraoperative blood loss and improve postoperative cognitive function is still inconclusive. So the investigators conduct the randomized control trial to compare the effect of magnesium with placebo control in blood loss and cognitive function in meningioma patient undergoing craniotomy.

DETAILED DESCRIPTION:
The investigators enroll 120 patient who admitted for craniotomy for meningioma removal. Then, the patients will be divided into two groups. The first group or group Mg will receive magnesium sulphate 40 mg/kg infuse for 30 min (started at skin incision), and then infuse magnesium sulphate 10 mg/kg/hr until the dura will be closed. The another group or normal saline group will receive the same amount of 0.9% sodium chloride. The anesthesia and surgery are standardized. The recorded data include patient demographic data, intraoperative blood loss, hemodynamics and pre and postoperative Montreal cognitive assessment score.

ELIGIBILITY:
Inclusion Criteria:

* Meningioma patient
* Schedule for supratentorial craniotomy with tumor removal
* American society of anesthesiologists physical status 1-3
* Age 18-70 years
* No alteration of conscious (full Glasgow coma score) and well cooperate
* Expected to extubation after operation

Exclusion Criteria:

* Unstable hemodynamic (severe hypotension or hypertension who receive antihypertensive and vasopressor before surgery but not include baseline oral antihypertensive drug)
* Known cardiac disease from either history, physical examination or investigation
* Patient who have heart block
* Hepatic disease (Child Pugh Score Class C)
* Renal insufficiency (eGFR < 60 ml/min from Chronic Kidney Disease Epidemiology Collaboration equation)
* Allergy to magnesium or other drugs use in the study
* Patient who receive calcium channel blocker drug
* Pregnancy
* Patient who receive magnesium for treatment such as arrhythmia or preeclampsia
* Hypermagnesemia (more than 2.6 mg/dL) before surgery
* BMI more than 30 kg/m2
* Patient who probably have brain herniation from increase intracranial pressure

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2020-02-03 (Actual); Study Completion 2020-02-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Manee Raksakietisak, M.D., Principal Investigator — Mahidol University
Locations (1):
- Faculty of medicine, Siriraj hospital, Mahidol University, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ostrom QT, Gittleman H, Farah P, Ondracek A, Chen Y, Wolinsky Y, Stroup NE, Kruchko C, Barnholtz-Sloan JS. CBTRUS statistical report: Primary brain and central nervous system tumors diagnosed in the United States in 2006-2010. Neuro Oncol. 2013 Nov;15 Suppl 2(Suppl 2):ii1-56. doi: 10.1093/neuonc/not151. No abstract available. PMID 24137015
- [Background] Wiemels J, Wrensch M, Claus EB. Epidemiology and etiology of meningioma. J Neurooncol. 2010 Sep;99(3):307-14. doi: 10.1007/s11060-010-0386-3. Epub 2010 Sep 7. PMID 20821343
- [Background] Goldbrunner R, Minniti G, Preusser M, Jenkinson MD, Sallabanda K, Houdart E, von Deimling A, Stavrinou P, Lefranc F, Lund-Johansen M, Moyal EC, Brandsma D, Henriksson R, Soffietti R, Weller M. EANO guidelines for the diagnosis and treatment of meningiomas. Lancet Oncol. 2016 Sep;17(9):e383-91. doi: 10.1016/S1470-2045(16)30321-7. Epub 2016 Aug 30. PMID 27599143
- [Background] Hooda B, Chouhan RS, Rath GP, Bithal PK, Suri A, Lamsal R. Effect of tranexamic acid on intraoperative blood loss and transfusion requirements in patients undergoing excision of intracranial meningioma. J Clin Neurosci. 2017 Jul;41:132-138. doi: 10.1016/j.jocn.2017.02.053. Epub 2017 Mar 7. PMID 28283245
- [Background] Soliman R, Fouad E. The effects of dexmedetomidine and magnesium sulphate in adult patients undergoing endoscopic transnasal transsphenoidal resection of pituitary adenoma: A double-blind randomised study. Indian J Anaesth. 2017 May;61(5):410-417. doi: 10.4103/ija.IJA_581_16. PMID 28584351
- [Background] Kutlesic MS, Kutlesic RM, Mostic-Ilic T. Magnesium in obstetric anesthesia and intensive care. J Anesth. 2017 Feb;31(1):127-139. doi: 10.1007/s00540-016-2257-3. Epub 2016 Nov 1. PMID 27803982
- [Background] Herroeder S, Schonherr ME, De Hert SG, Hollmann MW. Magnesium--essentials for anesthesiologists. Anesthesiology. 2011 Apr;114(4):971-93. doi: 10.1097/ALN.0b013e318210483d. PMID 21364460
- [Background] Rodriguez-Rubio L, Nava E, Del Pozo JSG, Jordan J. Influence of the perioperative administration of magnesium sulfate on the total dose of anesthetics during general anesthesia. A systematic review and meta-analysis. J Clin Anesth. 2017 Jun;39:129-138. doi: 10.1016/j.jclinane.2017.03.038. Epub 2017 Apr 7. PMID 28494889
- [Background] Modanlou Juibari H, Eftekharian HR, Arabion HR. Intravenous Magnesium Sulfate to Deliberate Hypotension and Bleeding after Bimaxillary Orthognathic Surgery; A Randomized Double-blind Controlled Trial. J Dent (Shiraz). 2016 Sep;17(3 Suppl):276-282. PMID 27840841
- [Background] Ghodraty MR, Homaee MM, Farazmehr K, Nikzad-Jamnani AR, Soleymani-Dodaran M, Pournajafian AR, Nader ND. Comparative induction of controlled circulation by magnesium and remifentanil in spine surgery. World J Orthop. 2014 Jan 18;5(1):51-6. doi: 10.5312/wjo.v5.i1.51. eCollection 2014 Jan 18. PMID 24649414
- [Background] Srivastava VK, Mishra A, Agrawal S, Kumar S, Sharma S, Kumar R. Comparative Evaluation of Dexmedetomidine and Magnesium Sulphate on Propofol Consumption, Haemodynamics and Postoperative Recovery in Spine Surgery: A Prospective, Randomized, Placebo Controlled, Double-blind Study. Adv Pharm Bull. 2016 Mar;6(1):75-81. doi: 10.15171/apb.2016.012. Epub 2016 Mar 17. PMID 27123421
- [Background] Elsharnouby NM, Elsharnouby MM. Magnesium sulphate as a technique of hypotensive anaesthesia. Br J Anaesth. 2006 Jun;96(6):727-31. doi: 10.1093/bja/ael085. Epub 2006 May 2. PMID 16670112
- [Background] Mack WJ, Kellner CP, Sahlein DH, Ducruet AF, Kim GH, Mocco J, Zurica J, Komotar RJ, Haque R, Sciacca R, Quest DO, Solomon RA, Connolly ES, Heyer EJ. Intraoperative magnesium infusion during carotid endarterectomy: a double-blind placebo-controlled trial. J Neurosurg. 2009 May;110(5):961-7. doi: 10.3171/2008.9.17671. PMID 19199498
- [Background] Bilotta F, Gelb AW, Stazi E, Titi L, Paoloni FP, Rosa G. Pharmacological perioperative brain neuroprotection: a qualitative review of randomized clinical trials. Br J Anaesth. 2013 Jun;110 Suppl 1:i113-20. doi: 10.1093/bja/aet059. Epub 2013 Apr 5. PMID 23562933
- [Background] Mathew JP, White WD, Schinderle DB, Podgoreanu MV, Berger M, Milano CA, Laskowitz DT, Stafford-Smith M, Blumenthal JA, Newman MF; Neurologic Outcome Research Group (NORG) of The Duke Heart Center. Intraoperative magnesium administration does not improve neurocognitive function after cardiac surgery. Stroke. 2013 Dec;44(12):3407-13. doi: 10.1161/STROKEAHA.113.002703. Epub 2013 Oct 8. PMID 24105697
- [Background] Mirrahimi B, Mortazavi A, Nouri M, Ketabchi E, Amirjamshidi A, Ashouri A, Khajavi M, Mojtahedzadeh M. Effect of magnesium on functional outcome and paraclinical parameters of patients undergoing supratentorial craniotomy for brain tumors: a randomized controlled trial. Acta Neurochir (Wien). 2015 Jun;157(6):985-91; discussion 991. doi: 10.1007/s00701-015-2376-x. Epub 2015 Apr 1. PMID 25824556
- [Background] Yang L, Wang HH, Wei FS, Ma LX. Evaluation of acute normovolemic hemodilution in patients undergoing intracranial meningioma resection: A quasi-experimental trial. Medicine (Baltimore). 2017 Sep;96(38):e8093. doi: 10.1097/MD.0000000000008093. PMID 28930850

RESULTS

PARTICIPANT FLOW:
Groups:
- Group NSS: The patients received normal saline with the same amount of magnesium sulphate for loading and continuous infusion started at skin incision until dura was closure. Anesthesia was maintained with propofol, fentanyl, cisatracurium and sevoflurane. Vasopressor or antihypertensive drug are used to control hemodynamics.
- Group Mg: The patients received 40 mg/kg of magnesium sulphate loading in 30 minutes at incision and then continuous drip 10 mg/kg/hr until dura was closure. Anesthesia was maintained with propofol, fentanyl, cisatracurium and sevoflurane. Vasopressor or antihypertensive drug are used to control hemodynamics.
Period: Overall Study
Arm/Group | Group NSS | Group Mg
Started | 40 | 40
Completed | 38 | 38
Not Completed | 2 | 2
Not completed — Protocol Violation | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group NSS | Group Mg | Total
Number analyzed (Participants) | 38 | 38 | 76
Age, Continuous [Mean (Standard Deviation); unit: years] | 52 (9.6) | 47 (11) | 50 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 34 | 68
  Male | 4 | 4 | 8
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 23.8 (3.6) | 23.3 (3.2) | 23.6 (3.4)
American Society of Anesthesiologist (ASA) [Count of Participants; unit: Participants] — ASA I is normal healthy patient ASI II is a patient with mild systemic disease such obesity (BMI > 30), well controlled hypertension, well controlled DM, mild lung disease
  Participants
    ASA I | 25 | 22 | 47
    ASA II | 13 | 16 | 29
Hemoglobin [Mean (Standard Deviation); unit: g/dL] | 13 (1.5) | 13 (1.2) | 13 (1.4)
Baseline mean arterial pressure [Mean (Standard Deviation); unit: mmHg] | 95 (12) | 93 (10) | 94 (11)
Single/multiple tumor [Count of Participants; unit: Participants]
  Single | 34 | 33 | 67
  Multiple | 4 | 5 | 9
Re-craniotomy [Count of Participants; unit: Participants] | 8 | 10 | 18
Baseline MOCA scores [Median (Full Range); unit: score on the MOCA scale] — MOCA or Montreal Cognitive Assessment is a screening instrument used to facilitate the assessment of cognitive impairment.
  MOCA scores range between 0-30, do higher values represent a better outcome. A score of 26 or over is considered to be normal.
  score on the MOCA scale | 21 [14 to 28] | 23 [11 to 28] | 22 [11 to 28]

OUTCOME MEASURES:

1. Primary Outcome: Intraoperative Blood Loss
Description: We measure the amount of blood loss in the operative room in suction box, gauze and plastic bag. The unit measure is millimeter.
Time Frame: Intraoperative period from skin was incised to the skin was closure, an average 5 hours.
Measure: Median (Full Range); unit: ml
Arm/Group | Group NSS | Group Mg
Number analyzed (Participants) | 38 | 38
ml | 510 [100 to 1600] | 500 [70 to 2300]
Statistical Analysis 1: Comparison: Group NSS vs Group Mg; Test type: Superiority; p = 0.315, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Intraoperative Packed Red Cell (PRC) Transfusion
Description: The amount of blood transfusion in patient who required PRC transfusion intraoperatively.
Time Frame: Intraoperative period from skin was incised to the skin was closure, an average 5 hours.
Measure: Median (Full Range); unit: unit of packed red cell
Arm/Group | Group NSS | Group Mg
Number analyzed (Participants) | 38 | 38
unit of packed red cell | 2 [1 to 4] | 1 [1 to 3]
Statistical Analysis 1: Comparison: Group NSS vs Group Mg; Test type: Superiority; p = 0.270, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Postoperative MOCA Score
Description: MOCA or Montreal Cognitive Assessment is a screening instrument used to facilitate the assessment of cognitive impairment.
  MOCA scores range between 0-30, do higher values represent a better outcome. A score of 26 or over is considered to be normal. We measure Montreal assessment score for assess cognitive function after operation at postoperative day 3-7.
Time Frame: Postoperative day 3-7
Population: There are some missing data due to patient's visual, hearing or writing problems that occurred postoperatively.
Measure: Median (Full Range); unit: score on the MOCA scale
Arm/Group | Group NSS | Group Mg
Number analyzed (Participants) | 15 | 16
score on the MOCA scale | 23 [15 to 28] | 25 [8 to 30]
Statistical Analysis 1: Comparison: Group NSS vs Group Mg; Test type: Superiority; p = 0.299, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Sevoflurane Requirement
Description: Amount of sevoflurane agents usage during surgery. The unit of measurement of volatile agent is minimum alveolar concentration (MAC). 1 MAC-hour was defined as 2% of sevoflurane for 1 hour duration.
Time Frame: Intraoperative period from skin was incised to the skin was closure, an average 5 hours.
Measure: Mean (Standard Error); unit: average minimum alveolar concentration
Arm/Group | Group NSS | Group Mg
Number analyzed (Participants) | 38 | 38
average minimum alveolar concentration | 0.65 (0.12) | 0.66 (0.17)

5. Secondary Outcome: Fentanyl Requirement
Description: Amount of fentanyl usage during surgery
Time Frame: Intraoperative period from skin was incised to the skin was closure, an average 5 hours.
Measure: Mean (Standard Error); unit: mcg/kg/hr
Arm/Group | Group NSS | Group Mg
Number analyzed (Participants) | 38 | 38
mcg/kg/hr | 0.65 (0.19) | 0.6 (0.18)

6. Secondary Outcome: Cis-atracurium Requirement
Description: Amount of cis-atracurium usage during surgery
Time Frame: Intraoperative period from skin was incised to the skin was closure, an average 5 hours.
Measure: Mean (Standard Error); unit: mg/kg/hr
Arm/Group | Group NSS | Group Mg
Number analyzed (Participants) | 38 | 38
mg/kg/hr | 0.08 (0.02) | 0.08 (0.01)

7. Secondary Outcome: Patient Received Intraoperative Packed Red Cell (PRC)
Description: Number of patients who required Intraoperative PRC transfusion
Time Frame: Intraoperative period from skin was incised to the skin was closure, an average 5 hours.
Measure: Count of Participants; unit: Participants
Arm/Group | Group NSS | Group Mg
Number analyzed (Participants) | 38 | 38
Participants | 10 | 7

ADVERSE EVENTS:
Time Frame: adverse event that occurred in the operating room until discharge from hospital, an average 8 days but maximum is 35 days
Arm/Group | Group NSS | Group Mg
All-Cause Mortality (participants affected / at risk) | 0/38 | 0/38
Serious Adverse Events (participants affected / at risk) | 1/38 | 1/38
Other Adverse Events (participants affected / at risk) | 17/38 | 13/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group NSS (N=38) | Group Mg (N=38)
Severe brain edema (Nervous system disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group NSS (N=38) | Group Mg (N=38)
Minor neurological complication (Nervous system disorders) | 10 | 12 — Seizure, CN palsy, Delirium, Hemiparesis, CSF leakage, Diabetes inspires (specific adverse event terms cannot be separated)
Infection (Infections and infestations) | 7 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-08-01): https://cdn.clinicaltrials.gov/large-docs/16/NCT03558516/Prot_000.pdf
  • Statistical Analysis Plan (2018-08-01): https://cdn.clinicaltrials.gov/large-docs/16/NCT03558516/SAP_001.pdf